CLINICAL TRIAL: NCT01954511
Title: Effects of Manual Therapy and Exercises Applied to Cervical Spine in Patients With Temporomandibular Disorders: Pilot Study
Brief Title: Manual Therapy and Exercises Applied to Cervical Spine in Patients With Temporomandibular Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was suspended for personal issues
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Bruno Leonardo da Silva Grüninger, Pt, Universidade Federal de Sao Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1139-4055; 0300.0.135.000-11 (Other: CEP/UFSCar)
Record Dates: First submitted 2013-09-17; First posted 2013-10-01 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome
Keywords: Stomatognathic diseases;; Temporomandibular Joint Dysfunction Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Stomatognathic Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manual therapy (No Intervention): Upper cervical flexion mobilization, C5 central posterior-anterior mobilization, Pressure biofeedback device
  Interventions: Other: Manual therapy; Device: Pressure biofeedback device

INTERVENTIONS:
Other: Manual therapy — The patient was supine with the cervical spine in a neutral position. The therapist brought about a contact of the occipital bone with the ﬁrst ﬁnger and medial aspect of the hand, and other hand over the frontal region of the patient's head. The mobilizing force was delivered by ﬂexing the upper cervical region using a combination of cephalic traction with the occipital hand and caudal pressure with the frontal hand. This technique was applied for 10 minutes
  Other Names: Upper cervical flexion mobilization
Other: Manual therapy — The patient was prone with the cervical spine in a neutral position. The therapist placed the tips of his thumbs on the posterior surface of the C5 spinous process, while the other ﬁngers rested gently around the patients' neck. This technique was applied for 9 minutes
  Other Names: C5 central posterior-anterior mobilization
Device: Pressure biofeedback device — Device: Stabilizer - Chattanooga Group Inc., Chattanooga, Tennessee, USA The cranio-cervical flexor stabilization exercise was done 10 times holding 10 seconds the flexing position graded through feedback from a pressure biofeedback device
  Other Names: Stabilizer

SUMMARY:
The objective of this study was to investigate the effect of a manual therapy and exercise program, focused on the rehabilitation of cervical function, on clinical signs and mandibular function in subjects with TMD.

DETAILED DESCRIPTION:
Temporomandibular disorder (TMD) is a general term that refers to disorders associated with the temporomandibular joint (TMJ) and the masticatory muscles. Among the main symptoms are pre-auricular pain (in the region of the TMJ) and/or pain in the masticatory muscles.

It's usual to observe that subjects with TMD also present cervical alteration. Beside this, cervical postural alterations produced by muscle tension can influence mandibular position.

The intervention protocol was based on manual therapy, stabilization exercises and stretching.

The technique are:.

1. Upper cervical flexion mobilization;
2. C5 central posterior-anterior mobilization;
3. Stabilization exercise: Cranio-cervical flexor stabilization exercise
4. Stretching of muscles: upper trapezius, scalenes, semispinalis capitis; splenius capitis, sternocleidomastoid

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with myogenic or mixed temporomandibular disorders

Exclusion Criteria:

* Patients diagnosed with arthrogenic or discogenic temporomandibular disorders

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changing in maximum mouth opening pain free | Before and 5 days follow-up intervetion
  The clinical signs was based on Research Diagnostic Criteria protocol and it was measured maximum mouth opening pain free using a caliper ((Somet, 150mm, Inox, Czechoslovakia)

SECONDARY OUTCOMES:
Changing of Pain | Before and 5 days follow-up intervetion
  To evaluate pain it was applied a scale from Research Diagnostic Criteria protocol, that consists of a line scored from 0 to 10, where 0 represents no pain and 10 the worst pain that the subject has experienced, allowing it to check the number that features their pain at the moment.

OTHER OUTCOMES:
Changing in Mandibular Function Impairment Questionnaire -MFIQ | Before and 5 days follow-up intervetion
  To evaluated mandibular function was used the Mandibular Function Impairment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ana Beatriz Oliveira, Phd, Study Director — Clinical professor - UFSCar; Letícia Bojikian Calixtre, Pt, Principal Investigator — UFSCar; Francisco Alburquerque Sendín, Phd, Principal Investigator — University of Salamanca; Melina Nevoeiro Haik, MSc, Principal Investigator — UFSCar